CLINICAL TRIAL: NCT03752294
Title: A 24-month, Randomized-control, Double-blind, Multi-center, Delayed-start, Pilot Study Evaluating Thrombin Inhibitions Alzheimer's Disease Using 150mg Dabigatran Daily: A Novel Therapeutic Target for Alzheimer's Disease
Brief Title: A Novel Therapeutic Target for Alzheimer's Disease in Men and Women 50-85 Years of Age.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: University of Rhode Island (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN001-001
Record Dates: First submitted 2018-05-15; First posted 2018-11-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment; Mild Alzheimer's Disease
Keywords: MCI; Mild AD; Dabigatran
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dabigatran; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Randomized-control, Double-blind, Multicenter, Delayed-start, Pilot
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The first phase of the study is 9-month, double-blind, randomized-control treatment. All participants participants will cross-over to phase II (open label) for an additional 12 months of treatment with a 3-month non-treatment follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dabigatran (Active Comparator): Participants will receive 150mg dabigatran daily for a total of 9-months.
  Interventions: Drug: Dabigatran
- Placebo (Placebo Comparator): Participants will receive placebo daily for a total of 9-months.
  Interventions: Drug: Placebo - Cap
- Open Label (Active Comparator): All study participants are assigned to receive 150mg dabigatran daily for a total of 12 months (study month 9 through month 21)
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — At the end of a 9-month randomized-control, double-blind treatment all study participants will cross-over to the 12-month open-label phase with a 3-month non-treatment follow-up.
  Other Names: Pradaxa
  Arms: Dabigatran; Open Label
Drug: Placebo - Cap — At the end of a 9-month randomized-control, double-blind treatment all study participants will cross-over to the 12-month open-label phase with a 3-month non-treatment follow-up
  Other Names: Study Drug
  Arms: Placebo

SUMMARY:
A randomized-control, double-blind, multi-center, delayed-start, pilot trial evaluating the disease modifying effects of a 150mg once-a-day dose vs. placebo of dabigatran in men and women, between the ages of 50-85 years, confirmed with MCI probably due to AD and mild Alzheimer's Disease.

DETAILED DESCRIPTION:
The study will be conducted in 2-phases. The Phase I double-blind portion of the study consists of 40-60 active participants with MCI probably due to AD and mild AD randomized to 150mg once-a-day dose of dabigatran or placebo. A futility analysis will be conducted based on month 3 plasma biomarker changes from baseline. Excluding futility, at the end of Phase I, the study continues onto the open-label phase of the study where the placebo arm will be treated with 150mg once-a-day with dabigatran from months 10-21. The active treatment arm will continue on dabigatran through month-21. For final analysis, a difference in intercept of a generalized growth model between randomization groups during Phase 2 in the Cognitive Dementia Rating Scale-Sum of Boxes (CDR-SB) will be taken as evidence of effectiveness and justify further study. All patients will discontinue dabigatran after month 21 and a 3-month follow-up period will confirm whether or not the proposed cognitive effects can be sustained in the absence of treatment. The relationships between changes in levels of plasma biomarkers over time will be tested with regards to each other and relative to MRI and cognitive testing performed at scheduled intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MCI likely due to AD or mild AD based on IWG-2 criteria for typical AD (A plus B at any stage) 2011 revised criteria
2. English speaking men & woman age 50 -85 years (inclusive)
3. Ability to provide informed consent
4. MMSE score >20 at screening
5. Informant or caregiver (e.g. family member, friend) willing to participate in semi-structured interviews
6. CSF Aβ positive (MCI and AD) or a positive amyloid positron emission tomography (PET) scan within 6-months prior to screening using IWG-2 criteria.
7. CDR Scale Global Score between 0.5 and 1
8. Stable dosing (prior 3-months) of standard AD medications are allowed
9. Demonstrated willingness to comply with study visit schedule, laboratory studies, and other study procedures

Exclusion Criteria:

1. Pre-menopausal women (last menstruation < 1 year prior to screening) who are not surgically sterile.
2. Creatinine clearance < 50mL/min
3. Current psychiatric or neurological disorder that would contribute to cognitive impairment (focal neurological features early extrapyramidal signs, early hallucinations, cognitive fluctuations, non-AD dementia, major depression)
4. Cerebrovascular disease
5. Toxic, inflammatory, and metabolic disorders, all of which may require specific investigations
6. MRI Flair or T2 signal changes in the medial temporal lobe that are consistent with infectious or vascular insults
7. Sudden onset or early occurrence of the following symptoms: gait disturbances, seizures, major and prevalent behavioral changes
8. Inability to swallow pills
9. Current anticoagulant therapy
10. Conditions associated with an increased risk of bleeding (e.g. major surgery within 30-days of baseline, planned surgery or intervention during treatment period)
11. History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
12. Gastrointestinal hemorrhage within the past year
13. Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30-days; hemorrhagic disorder or bleeding diathesis
14. Need for anticoagulant treatment of disorders, fibrinolytic agents within 48-hours of study baseline, uncontrolled hypertension (systolic blood pressure greater than 180mm Hg and/or diastolic blood pressure greater than 100 mm Hg)
15. Recent malignancy or radiation therapy (within 6-months) and a survival rate of 3-years,
16. Active infective endocarditis
17. Active liver disease (including but not limited to persistent ALT, AST, Alk Phos greater than twice the upper limit of the normal range; active hepatitis C (positive HCV RNA)
18. Active hepatitis B (HBs antigen +, anti HBc IgM +), active hepatitis A
19. HIV/AIDS diagnosis

MRI exclusionary criteria

1. Brain Aneurysm Clip
2. Implanted neural stimulator
3. Implanted cardiac pacemaker or defibrillator
4. Cochlear implant
5. Ocular foreign body (e.g. metal shavings)
6. Other implanted medical devices: (e.g. Swan Ganz catheter, mechanical prosthetic heart)
7. Insulin pump
8. Metal shrapnel or bullet

Additional concomitant drug exclusionary criteria will be applied by investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate dabigatran efficacy in MCI and mild AD population using changes in targeted plasma and CSF biomarker levels at 9 and 21 months | 9 and 21-months
  Evaluate effectiveness of dabigatran (150mg daily) on disease modification measured by changes in targeted plasma and CSF biomarkers associated with the early stages of Alzheimer's disease

SECONDARY OUTCOMES:
Demonstrate a reduction in decline of cognitive function related to physical functioning in placebo arm after crossing over to 12-months of active treatment | 12 - 24 months
  Demonstrate an observed benefit of cognitive performance/function using the ADCS ADL MCI
Changes in cognitive performance in placebo arm after cross-over to open-label treatment phase | 24-months
  Evaluate effectiveness of dabigatran (150mg daily) using the CDR-SB
Safety and tolerability of dabigatran in experimental population (MCI and mild AD populations) based on reported serious and adverse events | 21-months
  Determine the safety and tolerability of dabigatran in MCI probably due to AD and mild AD population using physician and patient reported adverse events.
Evaluation of cognitive performance in placebo arm after cross-over to open-label treatment phase | 24-months
  Evaluate effectiveness of dabigatran (150mg daily) using the MoCA

CONTACTS AND LOCATIONS:
Overall Officials: Paula Grammas, PhD, Study Director — Executive Director of the Ryan Institute for Neuroscience; John Stoukides, MD, Principal Investigator — Medical Director, Rhode Island Mood & Memory Research Institute

IPD SHARING:
Plan to Share IPD: Undecided